CLINICAL TRIAL: NCT05914870
Title: Effects of Multicomponent Training Versus Cardiovascular Training as a Treatment for Hypertension in Adult Subjects
Acronym: ETTH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Noelia González-Gálvez, Principal Investigator, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UCMurcia-ETTH
Record Dates: First submitted 2023-06-05; First posted 2023-06-22 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Hypertension
Keywords: Hypertension; High Blood Pressure; Training Program; Multicomponent Exercise; Combined Exercise; Cardiovascular Exercise
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Multi-component training (Experimental): The Multicomponent Training programme will apply two main training units per session per day.
  This experimental group will perform 2 intervention sessions per week with a duration of 60 minutes each; 10 minutes for the preparatory phase to exercise in which they will perform joint mobility exercises and dynamic stretching; 40 minutes will be dedicated to the main phase of the training, 20 minutes for strength work, with two exercises, one for the upper body and one for the lower body, and 20 minutes for cardiovascular work; finally, 10 minutes for the post-exercise phase in which they will perform a return to calm and static stretching.
  The duration of the programme will be 12 weeks (3 months).
  Interventions: Other: Multi-component training
- Continuous Cardiovascular Training (Experimental): The Continuous Cardiovascular Training programme will apply a single main training unit per session per day.
  This experimental group will perform 2 intervention sessions per week with a duration of 60 minutes each; 10 minutes for the preparatory phase to exercise in which they will perform joint mobility exercises and dynamic stretching; 40 minutes for the main phase of the training where they will perform continuous aerobic work without changes in intensity during the session; finally, 10 minutes for the post-exercise phase in which they will perform a return to calm and static stretching.
  The duration of the programme is 12 weeks (3 months).
  Interventions: Other: Continuous Cardiovascular Training
- Control Group (No Intervention): The control group will not perform any physical exercise programme and will continue with their daily tasks.

INTERVENTIONS:
Other: Multi-component training — The multicomponent training group will perform 60 minutes of training per session:
  * 10 minutes of joint mobility exercises and dynamic stretching.
  * 20 minutes of strength work with 2 exercises; the first, bench press, at an intensity of 50% of your 1RM. The number of repetitions will be individualised for each subject by testing the loss of speed in the series with respect to the first repetition (15% loss); the second, the squat, at an intensity of 60% of your 1RM. The number of repetitions shall be individualised for each subject by means of the loss of speed test in the series with respect to the first repetition (10% loss). The rest between sets will be 3 minutes.
  * 20 minutes of continuous cardiovascular work. The intensity will be increased every 4 weeks, from week 1 to 4 between 55%-65%FCR or VO2peak, from week 5 to 8 between 65%-%75%FCR or VO2peak and from week 9 to 12 between 75%-%85%FCR or VO2peak.
  * 10 minutes of cool down and static stretching.
  Arms: Multi-component training
Other: Continuous Cardiovascular Training — The Continuous Cardiovascular Training group will perform 60 minutes of training per session distributed as follows:
  Preparatory Phase: 10 minutes of standardised warm-up with joint mobility exercises and dynamic stretching.
  Main Training Phase:
  In this phase we will work 40 minutes of continuous aerobic exercise, maintaining the same intensity range throughout the session. We will increase the intensity every 4 weeks, from 1 to 4 you will work between 55%-65%FCR or VO2peak, from 5 to 8 between 65%-%75%FCR or VO2peak and from 9 to 12 between 75%-%85%FCR or VO2peak.
  Post-training phase: 10' cool down and static stretching.
  Arms: Continuous Cardiovascular Training

SUMMARY:
Hypertension is the most prevalent risk factor and the third leading cause of death worldwide, responsible for an increase in cardiac events. International guidelines on cardiology and hypertension recommend the practice of regular physical exercise for the control and treatment of this disease. The main objective of the study will be to determine the effect of a Multicomponent Training programme versus a Cardiovascular Training programme on blood pressure levels in hypertensive adults. The work methodology will consist of a controlled, randomised, longitudinal and prospective clinical trial, with several simultaneous study branches; on the one hand, the interventions with Multicomponent Training; on the other hand, the interventions with Cardiovascular Training; and, finally, a control group. The sample will be composed of 75 adult hypertensive subjects, including men and women, divided into groups of 25 people, two intervention groups and one control group. The inclusion criteria will be adult subjects, aged 40-65 years, with controlled arterial hypertension and sedentary. Exclusion criteria will be pregnant women and hypertensive patients with serious diseases that prevent the safe practice of physical exercise. The intervention will last 12 weeks and training will be 2 days per week, 60 minutes per session. The variables of the pre-post intervention study will be haemodynamic parameters; body composition, abdominal perimeter, general and manual strength, cardiorespiratory capacity, lipid profile and glucose.

DETAILED DESCRIPTION:
Cardiovascular disease is the leading cause of premature death worldwide and hypertension (HTN) is the most prevalent cardiovascular risk factor, being the third leading cause of death worldwide and responsible for an increased risk of heart disease, encephalopathy and kidney disease. HTN tops the list of serious non-communicable diseases, accounting for 10.4 million deaths per year. International guidelines on HTN recommend a diagnosis of HTN when a person's systolic blood pressure (SBP) in consultation is ≥140 mmHg and/or diastolic blood pressure (DBP) ≥90 mmHg, after several measurements (at least 3 every 1-2 minutes) on different days have been taken and recorded. Non-pharmacological interventions should be key to the control and treatment of HTN; these interventions involve changes in habits and behaviours in daily life, and it is here where the practice of regular physical exercise is decisive. The main objective of the study will be to analyse and compare the effect of a Multi-Component Training (MCT) programme versus a Continuous Cardiovascular Training (CVT) programme on BP levels in adult hypertensive subjects. The working methodology will consist of a controlled, randomised, longitudinal and prospective clinical trial, with several simultaneous study branches; on the one hand, the intervention with Multicomponent Training; on the other hand, the intervention Continuous Training and, finally, the control group. The recruitment of the sample will be done in collaboration with the primary health care centres in order to recruit a total of 75 adult hypertensive subjects between men and women who will be divided into three groups of 25 people each, two intervention groups and one control group. The inclusion criteria for participation in the clinical trial will be adult subjects, between 40 and 65 years of age, with controlled arterial hypertension and who do not do physical exercise or have not done so in the last 12 months. Exclusion criteria will be pregnant women and hypertensive patients with serious diseases that prevent the safe practice of physical exercise (unstable coronary artery disease, heart failure, renal failure, severe pulmonary hypertension, uncontrolled diabetes). The intervention will consist of two different training programmes, one with EMC and one with ECVC, for 12 weeks (3 months), with a frequency of 2 days a week and a duration of 60 minutes per session. During this period of time, the different phases of the design of the training programmes will be exhaustively defined, from the planning phase, with the anamnesis of the subject, through the periodisation phase, where the mesocycles, microcycles, training sessions and training units will be organised, the programming phase, controlling and manipulating the operative variables of frequency, volume, intensity and density, until reaching the last phase of the process, which will be the training prescription phase, with the work methodology and the selection of exercises. The EMC programme will involve applying two main intra-session and daily training units, a first part focused on strength work and a second part for cardiovascular training. This group will train 60 minutes per session, 10 minutes for the preparatory phase to exercise, 40 minutes for the main phase of the training, 20 minutes of strength work and 20 minutes of cardiovascular work, and finally 10 minutes for the post-exercise phase. The ECVC programme will involve a single main training unit per session per day; in this intervention the training will be exclusively cardiovascular. This group will train 60 minutes per session, 10 minutes for the preparatory phase to exercise, 40 minutes for the main phase of training and, finally, 10 minutes for the post-exercise phase. The study variables and the instruments for the assessment of these variables pre-post intervention will be systolic and diastolic blood pressure, mean arterial blood pressure, pulse pressure, double product and basal heart rate which will be measured with the BPBIO-750 sphygmomanometer; body composition analysis (weight, musculoskeletal mass, fat mass and visceral fat area) and phase angle will be analysed with the InBody 770; abdominal perimeter will be measured with a tape measure; manual strength will be assessed with a Baseline hydraulic dynamometer and upper and lower body strength will be measured through execution speed with a progressive load test, bench press and squat respectively, for the estimation of 1RM; cardiorespiratory capacity will be assessed with a clinical test on a cycloergometer; lipid profile values (cholesterol, HDL, LDL, triglycerides) and glucose will be obtained with a blood biochemistry.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 40-65 years
* Controlled high blood pressure
* Sedentary

Exclusion Criteria:

* Pregnant women
* Hypertensive patients with serious diseases that prevent safe physical activity

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2023-06-20 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-09-29 (Actual)

PRIMARY OUTCOMES:
Changes in Blood Pressure from baseline at week 12. | Two times. Baseline and 12 weeks later
  Blood pressure (sytolic blood pressure and diastolic blood pressure) shall be assessed using the BPBIO-750 blood pressure monitor in millimetres of mercury (mmHg). The subject should sit down 5 minutes before the measurement to relax, without talking, with the back well positioned and without crossing the legs. After the 5 minutes of rest, proceed with the two programmed BP measurements, leaving 3 minutes between the two measurements

SECONDARY OUTCOMES:
Changes in Mean Blood Pressure from baseline at week 12 | Two times. Baseline and 12 weeks later
  Mean Blood Pressure will be assessed by BPBIO-750 sphygmomanometer in millimetres of mercury (mmHg)
Changes in Pulse Pressure from baseline at week 12 | Two times. Baseline and 12 weeks later
  Pulse Pressure shall be assessed by BPBIO-750 sphygmomanometer in millimetres of mercury (mmHg).
Changes in Dual Product from baseline at week 12 | Two times. Baseline and 12 weeks later
  The Dual Product will be assessed using the BPBIO-750 sphygmomanometer in millimetres of mercury (mmHg).
Changes in Baseline Heart Rate from baseline at week 12 | Two times. Baseline and 12 weeks later
  Baseline heart rate shall be assessed by BPBIO-750 sphygmomanometer in millimetres of mercury (mmHg).
Changes in weight from baseline at 12 weeks. | Two times. Baseline and 12 weeks later
  Weight will be assessed by bioimpedance with the DSM-BIA Multifrequency Segmental Segmental Body Composition Analyser InBody 770. For the assessment, subjects will be informed that they must have spent at least 3 hours since the last meal and 30 minutes without drinking; not have drunk alcohol in the previous 48 hours; go to the toilet 30 minutes before weighing and not wear metal items in contact with the skin such as rings, bracelets or watches.
Changes in Skeletal Muscle Mass from baseline at week 12 | Two times. Baseline and 12 weeks later
  Skeletal Muscle Mass shall be assessed by bioimpedance with the DSM-BIA Multifrequency Segmental Segmental Body Composition Analyser InBody 770
Changes in Body Fat Mass from baseline at week 12 | Two times. Baseline and 12 weeks later
  Body Fat Mass will be assessed by bioimpedance with the DSM-BIA Multifrequency Segmental Segmental Body Composition Analyser InBody 770.
Changes in Body Mass Index from baseline at week 12 | Two times. Baseline and 12 weeks later].
  BMI will be assessed by bioimpedance with the DSM-BIA Multifrequency Segmental Body Composition Analyser InBody 770.
Changes in Body Fat Percentage from baseline at week 12 | Two times. Baseline and 12 weeks later
  Body Fat Percentage will be assessed by bioimpedance with the DSM-BIA Multifrequency Segmental Body Composition Analyser InBody 770.
Changes in Visceral Fat from baseline at week 12 | Two times. Baseline and 12 weeks later
  Visceral Fat will be assessed by bioimpedance with the InBody 770 DSM-BIA Multifrequency Segmental Segmental Body Composition Analyser.
Changes in Phase Angle from Baseline at week 12 | Two times. Baseline and 12 weeks later
  Phase Angle will be assessed by bioimpedance with the DSM-BIA Multifrequency Segmental Body Composition Analyser InBody 770.
Changes in Waist circumference from baseline at week 12 | Two times. Baseline and 12 weeks later
  Waist circumference will be assessed according to the ISAK protocol, using a tape measure and recorded in centimetres (cm). The subject should stand with feet together, arms crossed over the chest and abdomen relaxed; the measurement will be taken at the narrowest point of the waist, between the 10th rib and the iliac crest, the subject will be asked to lower the arms to the sides of the body and will be measured at the end of a normal exhalation.
Changes in Total Cholesterol from Baseline at week 12 | Two times. Baseline and 12 weeks later
  Total Cholesterol will be assessed by blood biochemistry. It will be recorded in milligrams decilitres (mg/dl). To perform the blood biochemistry the subject must have been fasting for at least 6 hours.
Changes in HDL from baseline at week 12 | Two times. Baseline and 12 weeks later
  High density lipoproteins will be assessed by blood biochemistry. To be recorded in milligrams decilitres (mg/dl).
Changes in LDL from baseline at one week | Two times. Baseline and 12 weeks later
  Low density lipoproteins will be assessed by blood biochemistry. To be recorded in milligrams decilitres (mg/dl).
Changes in Triglycerides from baseline at week 12 | Two times. Baseline and 12 weeks later
  Triglycerides shall be assessed by blood biochemistry. It shall be recorded in milligrams decilitres (mg/dl).
Changes in Glucose from baseline at week 12 | Two times. Baseline and 12 weeks later
  Glucose will be assessed by blood biochemistry. It will be recorded in milligrams decilitres (mg/dl).
Change in Manual Handgrip Strength from baseline at week 12 | Two times. Baseline and 12 weeks later
  Manual Handgrip Strength will be assessed using a Baseline hand-held hydraulic dynamometer. It shall be recorded in kilograms (kg). For the measurement, the subject should sit in the chair, with the back supported by the backrest, feet flat on the floor and with the right elbow flexed at 90º; place the wrist in a neutral position with the thumb upwards gripping the dynamometer; the subject should squeeze with the greatest possible force and pressure. The same shall be repeated with the left hand. Two measurements shall be made with both hands.
Changes in Upper Body Strength from Baseline at week 12 | Two times. Baseline and 12 weeks later
  Upper body strength will be assessed with a progressive load test through running speed. It will be recorded in metres per second (m/s). The test will be performed with a bench press to estimate the1RM. It will be recorded in kilograms.
Changes in Lower Body Strength from Baseline at week 12 | Two times. Baseline and 12 weeks later
  Lower body strength will be assessed with a progressive load test through running speed. It will be recorded in metres per second (m/s). The test will be performed with a squat to estimate 1RM. It will be recorded in kilograms.
Changes in Cardiorespiratory Capacity from baseline at week 12 | Two times. Baseline and 12 weeks later
  Cardiorespiratory fitness will be assessed with a clinical test on a cycloergometer. It will be a step test, 2 minutes each step. The first 2 minutes will be performed without load and from that moment the test will begin with 2 minutes at 50w. This will be increased by 25w every 2 minutes until the subject reaches voluntary fatigue. VO2peak will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Noelia G González-Gálvez, PhD., Murcia, Spain

IPD SHARING:
Plan to Share IPD: No